CLINICAL TRIAL: NCT01422629
Title: High Intensity Focused Ultrasound (HIFU) to Treat Breast Fibroadenoma: a Feasibility Study. A Multicentric, Open, Uncontrolled Study
Brief Title: High Intensity Focused Ultrasound (HIFU) to Treat Breast Fibroadenoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theraclion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HIFU/F/FA/Dec2010
Record Dates: First submitted 2011-08-18; First posted 2011-08-24 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Breast Fibroadenoma
Keywords: Breast Fibroadenoma; High Intensity Focused Ultrasound
MeSH Terms: conditions — Fibroadenoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- High Intensity Focused Ultrasound (HIFU) (Experimental)
  Interventions: Device: Ultrasonic ablation device

INTERVENTIONS:
Device: Ultrasonic ablation device — High Intensity focused ultrasound treatment
  Other Names: TH-One

SUMMARY:
This study is a multicentre, open, uncontrolled trial for the observation of histological changes in breast fibroadenoma following high intensity focused ultrasound (HIFU).

This study will be conducted in France in 20 patients with breast fibroadenoma with indication for a surgical resection. The patient will receive an HIFU treatment and 6 months after treatment, the need of the surgery is evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of breast fibroadenoma based on:Clinical examination, Ultrasound image and mammogram for women older than 35 years, and histology
* Fibroadenoma size superior at 1 cm at its largest dimension (measured by Ultrasound)

Exclusion Criteria:

* Patient pregnant or lactating
* Microcalcifications within the lesion at the mammogram.
* History of breast cancer or history of laser or radiation therapy to the target breast
* Breast implant in the target breast.
* Fibroadenoma not clearly visible on the ultrasound images (in B mode)
* Patient participating in other trials using drugs or devices

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
HIFU induced tissue necrosis assessed by histology of excised gland or reduction volume of fibroadenoma | 6 months after HIFU treatment

SECONDARY OUTCOMES:
Volume reduction of the fibroadenoma | 12 months after HIFU treatment
  reduction in volume at 2, 4, 6 and 12 months after HIFU session or total regression of the fibroadenoma evaluated with ultrasound just before surgery
- Pain score during the HIFU treatment evaluated by the Visual Analog Scale. | at treatment
Percentage of patients with Adverse events | at 12 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Loïc BOULANGER, MD, Principal Investigator — Hôpital Jeanne de Flandre, CHU de Lille - FRANCE
Locations (2):
- France (2):
  - Hôpital Jeanne de Flandre, CHU de Lille 2 Avenue Oscar Lambret, Lille
  - Hôpital Américain de Paris, Neuilly-sur-Seine